CLINICAL TRIAL: NCT06879431
Title: The Impact of Cognitive Behavioral Intervention On Postoperative Delirium In School-aged Children With Sleep Disorder Undergoing Congenital Heart Surgery: A Multicenter, Randomized Controlled Clinical Trial
Brief Title: Preoperative Sleep Intervention on Postoperative Delirium in School-aged Children Undergoing Congenital Heart Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yan Fuxia (Other)
Responsible Party: Sponsor-Investigator, Yan Fuxia, principal investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-2602
Record Dates: First submitted 2025-02-25; First posted 2025-03-17 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Delirium - Postoperative; Sleep Problems; Congenital Heart Disease (CHD)
MeSH Terms: conditions — Emergence Delirium; Parasomnias; Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT group (Experimental): The intervention group received a short intensive cognitive-behavioral therapy (CBT) intervention 7-14 days before surgery
  Interventions: Behavioral: cognitive-behavioral intervention
- control group (No Intervention): no intervention was imposed on the control group

INTERVENTIONS:
Behavioral: cognitive-behavioral intervention — After enrollment in the experimental group, the guardians were asked to fill out a sleep diary every day before surgery to self-report the children's sleep, and to wear a somatic movement recorder to monitor sleep (non-dominant arm) (wGT3x-BT accelerometer, ActiGraph) during the preoperative hospitalization period, except during surgery, and then to wear it to record the sleep-related parameters until 7 days after surgery or before discharge from the hospital.Preoperative daily cognitive-behavioral interventions (developmental trials were guided with WeChat applets), including cognitive change, sleep hygiene, sleep restriction, stimulus control, and relaxation training
  Arms: CBT group

SUMMARY:
This is a multicenter, randomized, controlled clinical trial aimed to determine whether preoperative sleep interventions could reduce the incidence of adverse outcomes, such as postoperative delirium, in sleep-disordered school-aged children undergoing congenital heart surgery. The study will include infants and toddlers undergoing elective cardiac surgery with sleep disorders, assessed by the Children's Sleep Habits Questionnaire (CSHQ). All participants will be randomly assigned to the intervention group and Controll group in a 1:1 ratio. The intervention group received a short intensive cognitive-behavioral intervention 7-14 days before surgery, and no intervention was imposed on the control group. The results of this study will provide suggestions for the prevention of delirium after cardiac surgery.

DETAILED DESCRIPTION:
The study will be carried out in Fuwai Hospital, Chinese Academy of Medical Sciences, Anzhen Hospital Affiliated to Capital Medical University, Fuwai Central China Cardiovascular Hospital, Fuwai Cardiovascular Hospital of Yunnan Province, and Children's Hospital Affiliated to Capital Institute of Pediatrics.

The research process is as follows: Conduct a routine assessment of sleep disorders for the children visiting the outpatient clinic. The guardians fill out the online Children's Sleep Habits Questionnaire. Fully inform the children with sleep disorders and their guardians of all the contents and procedures of this trial. After obtaining informed consent and signing the informed consent form, conduct a further assessment on the children to determine whether they meet the inclusion and exclusion criteria. All enrolled children and their guardians will receive preoperative education for congenital heart disease in the outpatient clinic. After stratification by research center, the random block is set to 4 - 6, the R will be used to randomly assign subjects to the experimental group and the control group at a 1:1 ratio. After randomization, the parents of children in the experimental group register for a WeChat mini-program, and the children receive cognitive-behavioral interventions every day before surgery. Guardians need to strictly implement and cooperate with researchers through phone calls (during the waiting period for admission) or face-to-face communication (during the preoperative hospitalization period). The control group does not receive any intervention and follows routine clinical practice. To better control the quality of interventions for children aged 6 - 12 in the experimental group, the daily implementation status of parents is counted for the degree of implementation (0 - 100%) in the WeChat mini-program. Guardians record the children's daily sleep diaries (online questionnaires) before surgery. The day before surgery, parents fill out the online Children's Sleep Habits Questionnaire again and compare the scores with the baseline scores. After admission, children wear actigraphs until the day of surgery and until discharge after surgery to automatically record sleep-related information. After the children are enrolled in the study, relevant researchers will supervise the implementation of cognitive-behavioral interventions for the children once a day before surgery to ensure that the actigraph device functions properly during hospitalization and remind guardians to record electronic sleep diaries until the night before surgery. Follow-up will be conducted within 7 days after surgery or before discharge to evaluate outcomes such as delirium and pain. The primary outcome is the incidence of postoperative delirium, and secondary outcomes include postoperative sleep quality, pain score, perioperative organ injury (including AKI, acute lung injury, and postoperative liver dysfunction), clinical recovery and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 0-36 months
2. Scheduled to undergo elective corrective surgery for congenital heart disease under cardiopulmonary bypass.
3. Sleep disorder assessed by Children's Sleep Habits Questionnaire (CSHQ) (CSHQ score >48)

Exclusion Criteria:

1. Preoperative use of sleep therapy-related medications
2. The risk adjustment in congenital heart surgery-1 (RACHS-1 classification) ≥4
3. History of preoperative cardiac assist device, mechanical ventilation support, or asphyxia rescue
4. Emergency surgery or preoperative ICU admission
5. History of neurodevelopmental disorders such as autism spectrum disorder, attention deficit hyperactivity disorder, or psychiatric disorders such as depression
6. Combined severe hepatic and renal dysfunction
7. Combination of non-cardiac malformations (adenoid hypertrophy, tracheobronchial stenosis, polysplenism, anaplastic syndrome, Down syndrome, DiGeoge syndrome, diabetes mellitus, reproductive system abnormalities, anal atresia and Williams syndrome, eye disorders)
8. History of preoperative cerebral ischemia and hypoxia
9. Concurrent participation in other clinical trials
10. Refusal of the family to sign the informed consent form or poor compliance by the child

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 544 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative delirium | Postoperative 7 days

SECONDARY OUTCOMES:
Mechanistic endpoint: Concentration of plasma S-100β protein | Before surgery, at the end of surgery and 24 hours after surgery
  S-100β protein was used as a surrogate biomarker for the disruption of the blood-brain barrier.
Pain defined by the Wong-Baker faces pain scale (revision) | Postoperative 7 days
  The Faces Pain Scale-Revised (FPS-R) requires patients to rate their overall pain intensity on a scale from 0 (no pain) to 10 (worst possible pain). Simultaneously, the FPS-R provides six cartoon illustrations of facial expressions (ranging from smiling, sad, to agonized crying) to visually represent the pain levels corresponding to different score ranges. This design aligns with children's concrete thinking characteristics. During assessment, the child simply points to the numerical rating or cartoon face that best matches their perceived pain intensity, making it particularly suitable for children aged 4 to 12 years.
The incidence of postoperative Acute kidney injury | Within postoperative 7 days
The incidence of Pulmonary complication | Postoperative 7 days
The incidence of postoperative Liver dysfunction | Postoperative 7 days
Concentration of intestinal fatty acid binding protein (I-FABP) | before surgery, at the end of surgery and 24 hours after surgery
  one of markers of intestinal injury
Concentration of zonulin | before surgery, at the end of surgery and 24 hours after surgery
  One of markers of intestinal injury
Concentration of lipopolysaccharide (LPS) | before surgery, at the end of surgery and 24 hours after surgery
  one of markers of intestinal injury
Concentration of lipopolysaccharide binding protein (LBP) | before surgery, at the end of surgery and 24 hours after surgery
  One of markers of intestinal injury
Types and dosages of drugs used for postoperative sedation and analgesia | Postoperative 7 days or before discharge
Concentration of IL-6 | before surgery, at the end of surgery and 24 hours after surgery
Concentration of TNF-α | before surgery, at the end of surgery and 24 hours after surgery
Concentration of IL-1β | before surgery, at the end of surgery and 24 hours after surgery
Concentration of IFN-γ | before surgery, at the end of surgery and 24 hours after surgery
Concentration of IL-17 | before surgery, at the end of surgery and 24 hours after surgery
Concentration of C-reactive protein | before surgery, at the end of surgery and 24 hours after surgery
The duration of postoperative mechanical ventilation | From the end of the surgery to the removal of the tracheal intubation，up to 30days
The length of intensive care unit stay | From the end of the surgery to discharge from the hospital,up to 30 days
  The time spent in the intensive care unit.
The length of postoperative hospital stay | From the end of the surgery to the day of discharge from the hospital,up to 30 days
Average daily cost | admission to discharge, up to 30days
  total hospitalization cost divided by total length of stay

OTHER OUTCOMES:
Long-term Sleep quality score | 30 days, six months, 1 year postoperatively
  guardians scored sleep quality 1-5 using a sleep diary
Strengths and Difficulties Questionnaire Score | 6 months and 1 year after surgery
  The Strengths and Difficulties Questionnaire (SDQ) consists of 25 items (0-50 scores) assessing five main domains: emotional symptoms, behavioral problems, oppositional behaviors, peer relationship problems, and social competence. These dimensions allow researchers to get a comprehensive picture of a child's emotional and behavioral status, with higher scores being more severe. Guardians will be required to complete the electronic SDQ Parent Version Questionnaire at 6 months postoperatively and 1 year postoperatively
Readmission rate | 30 days,6 months,1 year after discharge
  the rate at which a patient is readmitted to the hospital for the same or a different health problem within 30 days/six months/1 year after discharge
1-year mortality | 1 year after surgery
  the death rate of 1 year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Fuxia Yan, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, China

IPD SHARING:
Plan to Share IPD: No